CLINICAL TRIAL: NCT00003671
Title: Protocol for Patients With Newly Diagnosed Better Risk Acute Lymphoblastic Leukemia (ALL): A POG Pilot Study
Brief Title: Combination Chemotherapy in Treating Children With Newly Diagnosed Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9705; POG-9705 (Other: Pediatric Oncology Group); CDR0000066768 (Other: Clinical Trials.gov)
Record Dates: First submitted 1999-11-01; First posted 2004-09-13 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Leukemia
Keywords: untreated childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; Leucovorin; Mercaptopurine; Methotrexate; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy Treatment (Experimental): See detailed description.
  Interventions: Drug: asparaginase; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: thioguanine; Drug: vincristine sulfate

INTERVENTIONS:
Drug: asparaginase
  Other Names: E. coli; Elspar; NSC #109229
Drug: cyclophosphamide
  Other Names: CTX; Cytoxan; NSC #026271; IND #7089
Drug: cytarabine
  Other Names: cytosine arabinoside; Ara-C; Cytosar; NSC #063878
Drug: daunorubicin hydrochloride
  Other Names: daunomycin; DNR; Cerubidine; NSC #82151
Drug: dexamethasone
  Other Names: Decadron; NSC #034521
Drug: leucovorin calcium
  Other Names: LCV; Wellcovorin; citrovorum factor; folinic acid; NSC #003590
Drug: mercaptopurine
  Other Names: 6-MP; Purinethol; NSC #000755
Drug: methotrexate
  Other Names: MTX; amethopterin; NSC #000740; IND #4291
Drug: thioguanine
  Other Names: 6-thioguanine; 6-TG; NSC #752
Drug: vincristine sulfate
  Other Names: VCR; Oncovin; NSC #067574; IND #7161

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating children who have newly diagnosed acute lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether a delayed multidrug intensification can be given in conjunction with methotrexate and leucovorin calcium rescue consolidation therapy in children with average risk acute lymphocytic leukemia. II. Determine the feasibility of delivering 6 courses of this therapy in these patients.

OUTLINE: This is a multicenter study. Induction: Patients receive oral dexamethasone twice daily on days 1-29, vincristine IV on days 1, 8, 15, and 22, and asparaginase intramuscularly (IM) on days 2, 5, 8, 12, 15, and 19. Patients receive methotrexate intrathecally (IT) on days 1 and 15. CNS 2 and 3 patients also receive methotrexate IT on days 8 and 22. Patients with M1 bone marrow receive oral mercaptopurine daily beginning on day 29. Patients with M2 bone marrow on day 29 receive oral dexamethasone twice daily on days 29-42, vincristine IV and daunorubicin IV over 15 minutes on days 29 and 36, and asparaginase IM on days 29, 32, 36, and 39. Patients with M3 bone marrow on day 29 or M2 or M3 bone marrow on day 43 are taken off study. Consolidation: Patients receive methotrexate IV over 4 hours once a week during weeks 7, 10, 13, 24, 27, and 30, oral leucovorin calcium every 6 hours for 5 doses beginning 42 hours after the start of methotrexate infusion, methotrexate IT during weeks 5, 9, 12, 16, 20, 21, and 29, asparaginase IM 3 times weekly during weeks 16 and 17, and oral mercaptopurine daily during weeks 5-14 and from week 24 until the end of consolidation. Patients receive oral dexamethasone twice daily during weeks 8, 16-18, and 28, vincristine IV on day 1 during weeks 8, 9, 16, 17, 18, 28, and 29, daunorubicin IV on day 1 during weeks 16, 17, and 18, cyclophosphamide IV over 30 minutes on day 1 during week 20, cytarabine IV or subcutaneously on days 2-5 during weeks 20 and 21, and oral thioguanine daily during weeks 20 and 21. Intensive continuation: Patients receive oral methotrexate every 6 hours for 24 hours during weeks 1, 3, 5, and 7, oral mercaptopurine daily, and oral leucovorin calcium every 12 hours for 1 day beginning 48 hours after the start of oral methotrexate. Patients also receive methotrexate IT during week 8, vincristine IV on day 1 during week 8, and oral dexamethasone twice daily for 7 days beginning with vincristine. Treatment repeats every 8 weeks for 6 courses. Another continuation: Patients receive oral methotrexate once weekly except during the week of methotrexate IT administration, oral mercaptopurine daily, methotrexate IT every 8 weeks, vincristine IV on day 1 during week 8, and oral dexamethasone twice daily for 7 days beginning with vincristine. Treatment continues for up to 130 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 months for 4 years and then annually for ten years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically newly diagnosed early B-cell or B-precursor or B-progenitor acute lymphocytic leukemia Prior registration on POG-9400, stratum 6 for induction therapy Average prognosis (neither very good nor very poor)

PATIENT CHARACTERISTICS: Age: Children Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: No prior therapy other than on POG-9400

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 1998-12; Primary Completion 2002-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Naomi J. Winick, MD, Study Chair — Simmons Cancer Center
Locations (57):
- United States (50):
  - Arizona Cancer Center, Tucson, Arizona
  - Lucile Packard Children's Hospital at Stanford, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Naval Medical Center - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Nemours Children's Clinic, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Walt Disney Memorial Cancer Institute, Orlando, Florida
  - St. Mary's Hospital, West Palm Beach, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Chicago, Illinois
  - Christ Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Via Christi Regional Medical Center-Saint Francis Campus, Wichita, Kansas
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Portland, Maine
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - St. John's Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - University of Missouri-Columbia Hospital and Clinics, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Oklahoma Memorial Hospital, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center, Tulsa, Oklahoma
  - James H. Quillen College of Medicine, Johnson City, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Medical School, Charleston Division, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier de L'Universite Laval, Sainte-Foy, Quebec
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- San Jorge Childrens Hospital, Santurce, Puerto Rico
- Clinique de Pediatrie, Geneva, Switzerland